CLINICAL TRIAL: NCT05635565
Title: Intensive Goal Training With Educational Strategies for Parents and Adolescents With Cerebral Palsy
Brief Title: Intensive Goal Training With Educational Strategies for Adolescents With Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federal University of Minas Gerais (Other)
Responsible Party: Principal Investigator, MARINA B BRANDAO, Adjunct professor, Federal University of Minas Gerais
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63692422.0.0000.5149
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial with 2 groups
Who Masked: Outcomes Assessor
Masking Description: The assessor will not have access to the group allocation of the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Individualized goal training (Active Comparator): This group will be submitted to individualized goal training, 3 hours/day, 5 times/week, over the course of two weeks, totaling 30 hours. Training will happen in a clinical setting. Adolescents will select their functional goals to be trained during the intervention period.
  Interventions: Other: Individualized goal training
- Individualized goal training with educational strategies (Experimental): This group will be submitted to individualized goal training with their caregivers, for 2 weeks, with 5 face-to-face meetings lasting 3 hours a day at the rehabilitation center. The other 5 meetings will be held online with the adolescent and their caregiver at the same time, via video communication platform. Adolescents will select their functional goals to be trained during the intervention period.
  Interventions: Other: Individualized goal training with educational strategies

INTERVENTIONS:
Other: Individualized goal training — This group will be submitted to individualized goal training, 3 hours/day, 5 times/week, over the course of two weeks, totaling 30 hours. Training will happen in a clinical setting. Adolescents will select their functional goals to be trained during the intervention period.
  Arms: Individualized goal training
Other: Individualized goal training with educational strategies — This group will be submitted to individualized goal training with their caregivers, for 2 weeks, with 5 face-to-face meetings lasting 3 hours a day at the rehabilitation center. The other 5 meetings will be held online with the adolescent and their caregiver at the same time, via video communication platform. Adolescents will select their functional goals to be trained during the intervention period.
  Arms: Individualized goal training with educational strategies

SUMMARY:
Adolescents with cerebral palsy (CP) have limitations to perform daily routine activities. The use of educational strategies associated to an approach based on motor learning principles was found to be effective in promoting motor outcomes in individuals with CP. The aim of the present study is to investigate the effectiveness of an intensive, goal-directed training associated with education for parents and adolescents in promoting the daily functioning of adolescents with CP. A randomized clinical trial, with 20 adolescents with CP, aged between 12 and 17 years and 11 months, and their respective caregivers. Adolescents will be randomly allocated into one of two groups: (a) intensive training of functional goals with adolescents or (b) intensive functional goal training with adolescents, including parenting and adolescent education strategies.

DETAILED DESCRIPTION:
Adolescents with cerebral palsy (CP) have limitations to perform daily routine activities. The use of educational strategies associated to an approach based on motor learning principles was found to be effective in promoting motor outcomes in individuals with CP. However, there is a shortage of services focused on the specific needs of adolescents with CP and on the skills considered important for the success of the transition period to adulthood. Complementarily, the literature reveals the scarcity of services that provide educational support to parents on how to deal with the functional limitations of their adolescent children with CP. Therefore, it is possible that the development of an intervention protocol that associates high intensity training with specific functional goals with an educational program for parents and adolescents, can contribute to the provision of rehabilitation services targeted at adolescents with CP and their families. The overall objective of the present study is to investigate the effectiveness of an intensive, goal-directed protocol associated with education for parents and adolescents in promoting the daily functioning of adolescents with CP. A randomized clinical trial will be conducted with 20 adolescents with CP, aged between 12 and 17 years and 11 months, and their respective caregivers. Adolescents will be randomly allocated into one of two groups: (a) intensive training of functional goals with adolescents (3 hours/day, 5 days/week, during two weeks, totaling 30 hours, in a clinical setting) or (b) intensive functional goal training with adolescents, including parenting and adolescent education strategies (3 hours/day, 5 days/week, during two weeks, totaling 30 hours, with telehealth strategies and visits at the clinical setting).

ELIGIBILITY:
Inclusion Criteria:

* Adolescents with: (a) medical diagnosis of CP (unilateral or bilateral); (b) age between 12 and 17 years and 11 months; (c) manual ability Classified by the Manual Ability Classification System - MACS, at levels I (adolescents capable of handling objects of effectively and independently) to III (adolescents with limited repertoire of activities, who handle objects with supervision or adaptation); (d) gross motor function classified by the Gross Motor Function Classification System - GMFCS Expanded and Revised (GMFCS E & R), in the levels I (adolescents who walk in different contexts, but have limited speed, balance and coordination to run and jump) to IV (adolescents who use a wheelchair in most contexts, but are able to sustain weight on their lower limbs to help in transfers and walking short distances with physical help from a person); (e) communication function classified by the Communication Function Classification System for Individuals with Cerebral Palsy (CFCS) at levels: I (communicates at a appropriate pace with little or no delay in understanding, elaborating a speech, or resolve a misunderstanding); II (independently alternates sender and receiver roles with most people in most situations, but the pace of conversation is slow).

Exclusion Criteria:

* Adolescents undergoing any type of intensive intervention, orthopedic surgery or application of botulinum toxin in the upper limbs and/or less than six months will be excluded.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Canadian Occupational Performance Measure (COPM) | 4 Months
  Canadian Occupational Performance Measure (COPM) - performance and satisfaction scales (each scale ranging 1-10; higher values, better outcomes)

SECONDARY OUTCOMES:
Pediatric Evaluation of Disability Inventory- Computer Adaptive Test | 4months
  The test is divided into four domains that assess adolescent's daily functioning: Daily Activities (AD), Mobility (MB), Social/Cognitive (SC) and Responsibility (RS). The AD, MB, and SC domains are scored on a scale of 1 (Unable, unable to manages) to 4 (Easy), whereas the RS domain the scale varies from 1 (adult assumes complete responsibility) to 5 (child/youth assumes full responsibility). Each domain has scaled scores, ranging from 0-100 (higher means that the participant has more functional abilities and responsibility).
Domains of Mastery Motivation (DMQ) - Self-reported | 4 months
  The self-reported version is developed for individuals from 13 to 19 years old . The questionnaire evaluates aspects of the perceptions of adults and adolescents about the domain of adolescents in challenging structured tasks.
  DMQ has 41 items and seven scales: (1) Persistence on objects or cognitive tasks; (2) Gross motor persistence; (3) Social domain motivation with adults (4) Social domain motivation; (5) Pleasure of mastery and (6) Negative reactions (failures) in situations of domain; (7) General competence. Participants will be asked to rate, on a five-point scale, points (from "not at all typical" to "very typical"), how typical is the behavior of the adolescents in each item. The total score is the index of motivation, with higher scores representing more level of overall motivation.
Domains of Mastery Motivation (DMQ) - Parent- report | 4 months
  The parent- report version is developed for parents of individuals from 13 to 19 years old . The questionnaire evaluates aspects of the perceptions of parents regarding their child's motivation in challenging tasks. DMQ has 41 items and seven scales: (1) Persistence on objects or cognitive tasks; (2) Gross motor persistence; (3) Social domain motivation with adults (4) Social domain motivation; (5) Pleasure of mastery and (6) Negative reactions (failures) in situations of domain; (7) General competence. Parents will be asked to rate, on a five-point scale, points (from "not at all typical" to "very typical"), how typical is the behavior of the adolescents in each item. The total score ( is the index of motivation, with higher scores representing more level of overall motivation, according to parents.
Depression, Anxiety and Stress Scales (DASS-21) | 4 months
  The DASS-21 will be conducted with parents. It is a set of three four-point Likert subscales, aimed at assessing the emotional states of depression, anxiety and stress. Each statement is answered by underlining how the person has felt during the last week. Answers are ranked on a scale from 0 to 3 and the result of each dimension is obtained by adding up the answers to the items in each subscale. The final score is the sum of the three sub-scales. The higher the score (0-63 points), the worst is the mental health condition.
Depression, Anxiety and Stress Scale for Adolescents (EDAE-A) | 4 months
  The EDAE-A will be conducted with adolescents.It is a set of three four-point Likert subscales, aimed at assessing the emotional states of depression, anxiety and stress. Each statement is answered by underlining how the person has felt during the last week. Answers are ranked on a scale from 0 to 3 and the result of each dimension is obtained by adding up the answers to the items in each subscale. The final score is the sum of the three sub-scales. The higher the score (0-63 points), the worst is the mental health condition.

CONTACTS AND LOCATIONS:
Locations (1):
- Marina de Brito Brandão, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Upon request, due to confidentiality issues.

REFERENCES:
- [Background] Feitosa AM, Mancini MC, Silverio APM, Gordon AM, Brandao MB. "Help Me to Improve my Own Priorities!": A Feasibility Study of an Individualized Intensive Goal Training for Adolescents with Cerebral Palsy. Phys Occup Ther Pediatr. 2021;41(6):601-619. doi: 10.1080/01942638.2021.1891186. Epub 2021 Mar 2. PMID 33653225